CLINICAL TRIAL: NCT04832555
Title: Non Elective Vulnerable Elderly Radiotherapy
Acronym: NEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Policlinico Modena (Other)
Responsible Party: Principal Investigator, Elisa D'angelo, Medical Doctor, MD, Azienda Ospedaliero Universitaria Policlinico Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEVER
Record Dates: First submitted 2021-03-05; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Elderly; Vulnerable; Radiotherapy; Non-elective Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open: non elective irradiation (Experimental): Patients within inclusion criteria will be enrolled in the experimental treatment: a radiation therapy addressed to non elective site of disease and with a simultaneous integrated boost
  Interventions: Radiation: Non elective radiotherapy

INTERVENTIONS:
Radiation: Non elective radiotherapy — Simultaneous integrated boost on CTV volumes, delineated as per guidelines, with the exception of intermediate-low risk, where the CTVs are experimental.

SUMMARY:
To evaluate whether patients defined "non-fit for curative non-surgical radio-chemotherapy" and therefore treated with RT alone addressed only to non-elective sites of disease, could obtain a non-inferior loco-regional control compared to similar historical cohorts.

DETAILED DESCRIPTION:
The current standard approach for head and neck malignancies cannot be considered the gold standard for elderly patients, except in carefully selected cases. Given the relevance of this population, scientific societies also suggest to propose prospective studies for this subset of frail patients (European Organization for Research and treatment of cancer (EORTC), European Society for Medical oncology (ESMO)). In addition, it is necessary to collect data on specific categories, which are as homogeneous as possible. Therefore, the purpose of this study is to evaluate efficacy and safety of a tailored RT approach administered with a curative intent in a subset of frails elderly patients not candidates neither to standard concurrent RT-CT / RT-cetuximab nor to palliative treatment/best supportive care.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced non-metastatic HNSCC patients older than 70 years
* Primary tumor clinically and radiologically detectable and measurable (staging according to ed. TNM VII and also VIII.
* patients defined by the tumor board (ENT, Oncologist, Radiotherapist, Nutritionist) as 1) not eligibles for RTCT / RT-cetuximab treatment 2) not amenable to radical surgery and 3) not candidates for treatments with palliative intent/best supportive care
* Availability of staging with CT/PET for distant metastasis and CT/MRI for primary tumor
* Karnofsky performance status (KPS) ≥60/100
* Oropharynx , Hypopharynx and Larynx, Oral cavity: stage III and IV and Unknown primitive P16-POSITIVE

Exclusion Criteria:

* Age less than 70 years

  * Staging exams done 45 days before the date of the beginning of the treatment
  * Subsites: nasopharynx, salivary glands, paranasal sinuses. Metastatic disease
  * Gross total excision
  * All subsites concerned if N3.
  * Squamous cell neoplasms of the glottic larynx T1-T2 N0.
  * Unknown primary HPV negative or EBV positive.
  * Presence of distant metastases or sub-clavicular lymphadenopathies.
  * Previous surgery on T and/or N except diagnostic tonsillectomy.
  * 3D-conformational radiotherapy technique

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Loco-regional control | 24 months after the start of treatment
  clinical or radiological (RECIST 1.1) disease progression from end of treatment with tumor present, or to the date of salvage surgery of primary tumor with tumor present performed for clinical or radiological (RECIST 1.1) disease progression, whichever comes first.

SECONDARY OUTCOMES:
rate of severe sub-acute or late toxicity | at 6 and 12 months after the completion of radiotherapy
  assessment of toxicity according to CTCAE v5.0 scale
Cause-specific mortality rates | within 3 months after start of treatment
  Patients who died from cancer/total amount
overall survival | 5 years
  defined as the time from the date of randomization to the date of death for any cause
progression free survival | 12 and 24 months
  per modified Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
G8 role | 6 and 12 months
  correlation between G8 pre-screening evaluation and toxicity

OTHER OUTCOMES:
radiomics | through study completion, an average of 5 year
  evaluation of radiomics features in study population: using an automated high-throughput extraction of large amounts of quantitative features

CONTACTS AND LOCATIONS:
Overall Officials: Elisa D'Angelo, Study Chair — Azienda Ospedaliero Universitaria Policlinico Modena
Locations (1):
- AOUPoliclinicoModena, Modena, Italy